CLINICAL TRIAL: NCT00634179
Title: A Phase I/II Trial of VR-CHOP for Patients With Untreated Follicular Lymphoma and Other Low Grade B-Cell Lymphomas
Brief Title: A Phase I/II Trial of VR-CHOP in Lymphoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Christopher R. Flowers, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00002996; X05215 (Other: Winship Cancer Institute)
Record Dates: First submitted 2008-02-11; First posted 2008-03-12 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-09

CONDITIONS: Lymphoma, B-Cell; Follicular Lymphoma
Keywords: Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma | interventions — Bortezomib; Rituximab; Doxorubicin; Cyclophosphamide; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (VR-CHOP regimen) (Experimental): INDUCTION: Patients receive bortezomib IV on days 1 and 8; rituximab IV, doxorubicin hydrochloride IV over 3-5 minutes, cyclophosphamide IV over 60 minutes, and vincristine sulfate IV over 10 minutes on day 1; and prednisone PO on days 1-5. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression.
  MAINTENANCE: Patients achieving complete response (CR) receive rituximab IV once every 12 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or partial response (PR) receive rituximab IV and bortezomib once weekly for 4 weeks every 6 months for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Biological: Rituximab; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Bortezomib — Bortezomib 1.6 mg/m² given on days 1 and 8
  Other Names: Velcade
Biological: Rituximab — Rituximab 375 mg/m²
  Other Names: Rituxin; MabThera
Drug: Doxorubicin — Doxorubicin 50 mg/m²
  Other Names: Adriamycin
Drug: Cyclophosphamide — Cyclophosphamide 750 mg/m²
  Other Names: Neosar
Drug: Vincristine — Vincristine 1.4 mg/m² (capped at 1.5 mg maximum) given on day 1
  Other Names: Oncovin
Drug: Prednisone — Prednisone 100 mg/day given orally on days 1-5
  Other Names: Deltasone

SUMMARY:
This is an open-label (doctors and patients know which drug will be given), single center, phase 1/2 clinical trial. The primary objective is to determine whether VR-CHOP provides benefit to patients with previously untreated indolent non-Hodgkin's lymphomas (NHL).

DETAILED DESCRIPTION:
This study will assess whether adding bortezomib (Velcade) to R-CHOP (in a new combination called VR-CHOP) can further improve outcomes in patients with indolent NHL who have not previously received treatment.

Patients who are eligible to take part in the study will receive VR-CHOP at the doses of Velcade and vincristine established in phase 1. Patients will receive VR-CHOP for up to 8 cycles of treatment (each of 21 days duration). During treatment, patients will be assessed for their response to therapy and for possible side effects. All patients will go on to receive maintenance therapy after completion of their initial treatment as designed by the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Tissue diagnosis of a previously untreated, cluster of differentiation antigen 20+ (CD20+), B-cell non-Hodgkin lymphoma.

  * For the Phase 1 trial: patients with any of the following diagnoses are eligible:

    * Follicular Lymphomas (Grade 1, 2, 3a, 3b)
    * Small Lymphocytic Lymphoma
    * Marginal Zone Lymphomas
  * For the Phase 2 trial: patients with any of the following diagnoses are eligible:

    * Follicular Lymphomas (Grade 1, 2, 3a)
    * Small Lymphocytic Lymphoma
    * Marginal Zone Lymphomas
* Patients with follicular or other low-grade lymphoma must have an indication for treatment based on modified Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria or a Follicular Lymphoma International Prognostic Index (FLIPI) score ≥ 3.

  * Indications for treatment based on modified GELF criteria include any one of the following:

    * B symptoms or other lymphoma-related symptoms
    * Involvement of 3 nodal sites, each with a diameter of 3 cm
    * Any nodal or extranodal tumor mass with a diameter of 7 cm
    * Splenomegaly greater than 16 cm by CT scan.
    * Pleural effusions or peritoneal ascites
    * Cytopenias (leukocytes < 1.0 x 10 /L and/or platelets < 100 x 10/L)
    * Leukemia (> 5.0 x 10 /L circulating malignant cells)
  * Indications for treatment based on FLIPI criteria include any three of the following:

    * Age ≥ 60 years
    * Ann Arbor stage III or IV
    * Hemoglobin level < 120 g/L
    * Number of nodal areas involved > 4
    * Serum lactate dehydrogenase (LDH) level > normal
* Only chemotherapy-naïve subjects are eligible. Subjects may have received prednisone (< 2 months of therapy) or radiation ≤ 2 sites of therapy.
* Voluntary written informed consent and Health Insurance Portability and Accountability Act (HIPAA) Authorization before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Female patients of child bearing potential must have a negative β-human chorionic gonadotropin (β-hCG) test.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* ≥ 18 years of age at the time of registration.
* Patients must have adequate renal function as demonstrated by a serum creatinine < 1.5 mg/dl unless felt to be secondary to lymphoma.
* Must have an alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 3.5 the upper limit of normal and a total bilirubin ≤ 2.0 mg/dL unless secondary to lymphoma.
* Must have a cardiac left ventricular ejection fraction ≥ 50%.
* At least 1 measurable tumor mass (greater than 1.5 cm in the longest dimension and greater than 1.0 cm in the short axis).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.

Exclusion Criteria:

* Subject with primary or secondary central nervous system (CNS) lymphoma (current or previously treated) will not be eligible.
* A history of unrelated (non-lymphomatous) neoplasm within the past 10 years other than non-melanoma skin cancer or in-situ cervix cancer. Subjects with a prior diagnosis of malignancy more than 10 years may be entered into the study at the discretion of the Principal Investigator.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patient has received other investigational drugs with 14 days before enrollment.
* Patient has hypersensitivity to boron or mannitol.
* Female subject is pregnant or breast-feeding. Chemotherapeutic agents are known to have teratogenic effects on developing embryos and to cause chromosomal damage to gametes. These agents also cause bone marrow suppression and can be excreted in milk. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has ≥ Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has a platelet count of < 10 x 10¹⁰/L (unless due to bone marrow involvement with lymphoma documented within 14 days before enrollment).
* Patient has an absolute neutrophil count of < 1.0 x 10⁹/L (unless due to bone marrow involvement with lymphoma documented within 14 days before enrollment).
* Patient has a calculated or measured creatinine clearance of < 20 mL/minute within 14 days before enrollment.
* Presence of antibodies to HIV.
* Subject unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Flowers, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Result] Sinha R, Kaufman JL, Khoury HJ Jr, King N, Shenoy PJ, Lewis C, Bumpers K, Hutchison-Rzepka A, Tighiouart M, Heffner LT, Lechowicz MJ, Lonial S, Flowers CR. A phase 1 dose escalation study of bortezomib combined with rituximab, cyclophosphamide, doxorubicin, modified vincristine, and prednisone for untreated follicular lymphoma and other low-grade B-cell lymphomas. Cancer. 2012 Jul 15;118(14):3538-48. doi: 10.1002/cncr.26660. Epub 2012 Jan 3. PMID 22535574
- [Result] Cohen JB, Switchenko JM, Koff JL, Sinha R, Kaufman JL, Khoury HJ, Bumpers N, Colbert A, Hutchison-Rzepka A, Nastoupil LJ, Heffner LT, Langston AA, Lechowicz MJ, Lonial S, Flowers CR. A phase II study of bortezomib added to rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone in patients with previously untreated indolent non-Hodgkin's lymphoma. Br J Haematol. 2015 Nov;171(4):539-46. doi: 10.1111/bjh.13637. Epub 2015 Aug 7. PMID 26248505

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited from Winship Cancer Institute of Emory University.
Pre-assignment Details: A total of 37 patients were enrolled. However, not all patients participated in both phases of this study. For phase I, 19 patients were enrolled, and for phase II, 30 patients were enrolled.
Groups:
- Treatment (VR-CHOP Regimen): Phase I will identify the maximal tolerated doses of bortezomib and vincristine when used in a combination of bortezomib, rituximab and the cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) chemotherapy regimen.
  In Phase II, the trial will evaluate the efficacy and safety of the MTD combination of VELCADE and rituximab-CHOP in additional subjects who have untreated follicular B-cell non-Hodgkin's lymphoma (B-NHL)(Grade 1, 2, 3a), small lymphocytic lymphoma, or marginal zone lymphoma.
Period: Phase I: Induction
Arm/Group | Treatment (VR-CHOP Regimen)
Started | 19
Completed | 19
Not Completed | 0
Period: Phase II: Maintenance
Arm/Group | Treatment (VR-CHOP Regimen)
Started | 30
Completed | 29
Not Completed | 1
Not completed — Diagnosis changed after re-review | 1

BASELINE CHARACTERISTICS:
Population: A total of 37 patients were enrolled on this study. However, not all patients participated in both phases of this study. For phase I, 19 patients were enrolled, and for phase II, 30 patients were enrolled.
Arm/Group | Treatment (VR-CHOP Regimen)
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 58 [28 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Maximal Tolerated Doses of Bortezomib and Vincristine When Used in Combination of Bortezomib, Rituximab and the CHOP Chemotherapy Regimen (Phase I)
Description: INDUCTION: Patients receive bortezomib IV on days 1 and 8; rituximab IV, doxorubicin hydrochloride IV over 3-5 minutes, cyclophosphamide IV over 60 minutes, and vincristine sulfate IV over 10 minutes on day 1; and prednisone PO on days 1-5. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression.
Time Frame: Cycle 1 for MTD, following completion of therapy for CR, up to 24 weeks
Measure: Number (95% Confidence Interval); unit: mg/m^2
Groups:
- MTD of Bortezomib With Vincristine Capped at 1.5 mg: Maximal tolerated dose (MTD) of bortezomib when vincristine is capped at 1.5 mg
Arm/Group | MTD of Bortezomib With Vincristine Capped at 1.5 mg
Number analyzed (Participants) | 19
mg/m^2 | 1.62 [0.63 to 1.88]

2. Secondary Outcome: An Estimate of the Overall Response Rate (ORR)(Complete Response [CR] + CR Unconfirmed [CRu] + Partial Response [PR]) to Bortezomib and Rituximab (VR)-CHOP According to International Workshop to Standardize Response Criteria (IWRC) Criteria
Description: Response was assessed by computerized tomography (CT) after every 2 cycles of induction therapy, one time at least 4 weeks after completing induction (i.e., prior to maintenance), and then every 3 months while on maintenance therapy. At the conclusion of maintenance therapy, patients underwent one post-treatment scan, with further scans completed at the discretion of the treating physician. Positron emission tomography was permitted but only CT measurements were used to determine response.
Time Frame: Following completion of therapy, up to 2 years
Measure: Number; unit: participants
Groups:
- Phase I: Induction: INDUCTION: Patients receive bortezomib IV on days 1 and 8; rituximab IV, doxorubicin hydrochloride IV over 3-5 minutes, cyclophosphamide IV over 60 minutes, and vincristine sulfate IV over 10 minutes on day 1; and prednisone PO on days 1-5. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression.
- Phase II: Maintenance: INDUCTION: Patients receive bortezomib IV on days 1 and 8; rituximab IV, doxorubicin hydrochloride IV over 3-5 minutes, cyclophosphamide IV over 60 minutes, and vincristine sulfate IV over 10 minutes on day 1; and prednisone PO on days 1-5. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression.
  MAINTENANCE: Patients achieving CR receive rituximab IV once every 12 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or PR receive rituximab IV and bortezomib once weekly for 4 weeks every 6 months for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Bortezomib: Bortezomib 1.6 mg/m² given on days 1 and 8
  Rituximab: Rituximab 375 mg/m²
  Doxorubicin: Doxorubicin 50 mg/m²
  Cyclophosphamide: Cyclophosphamide 750 mg/m²
  Vincristine: Vincristine 1.4 mg/m² (capped at 1.5 mg maximum) given on day 1
  Prednisone: Prednisone 100 mg/day given orally on
Arm/Group | Phase I: Induction | Phase II: Maintenance
Number analyzed (Participants) | 19 | 29
participants
  Complete Response (CR) | 13 | 19
  Partial Response (PR) | 6 | 10
  Overall Response Rate (ORR) | 19 | 29

ADVERSE EVENTS:
Groups:
- Phase I: Induction: Phase I will identify the maximal tolerated doses of bortezomib and vincristine when used in a combination of bortezomib, rituximab and the CHOP chemotherapy regimen.
- Phase II: Maintenance: In Phase II, the trial will evaluate the efficacy and safety of the MTD combination of VELCADE and rituximab-CHOP in additional subjects who have untreated follicular B-NHL. (Grade 1, 2, 3a), small lymphocytic lymphoma, or marginal zone lymphoma.
Arm/Group | Phase I: Induction | Phase II: Maintenance
Serious Adverse Events (participants affected / at risk) | 3/19 | 1/29
Other Adverse Events (participants affected / at risk) | 16/19 | 22/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Induction (N=19) | Phase II: Maintenance (N=29)
Thrombosis (Blood and lymphatic system disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Pain (Nervous system disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Anxiety/Depression (Psychiatric disorders) | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Extravasation (Blood and lymphatic system disorders) | 1 | 0
Prolonged QT Interval (Cardiac disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Induction (N=19) | Phase II: Maintenance (N=29)
Neutropenia (Blood and lymphatic system disorders) | 13 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 3
Nausea (General disorders) | 13 | 2
Neuropathy (Nervous system disorders) | 16 | 22
Fatigue (General disorders) | 11 | 1
Vomiting (Gastrointestinal disorders) | 9 | 2
Diarrhea (Gastrointestinal disorders) | 7 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Low Potassium (Metabolism and nutrition disorders) | 4 | 2
Pain (Nervous system disorders) | 12 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Extravasation (Blood and lymphatic system disorders) | 0 | 1
Fever (Immune system disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Parotitis (Immune system disorders) | 0 | 1
Weakness (General disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes